CLINICAL TRIAL: NCT00237263
Title: An Extension Study to Phase IIb Dose-finding Study of Entacapone in Patients With Parkinson's Disease With End-of-dose Wearing-off
Brief Title: An Extension Study of Entacapone in Patients With Parkinson's Disease With End-of-dose Wearing-off. This Study is Not Recruiting in the United States
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCOM998A1204
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease, end-of -dose wearing-off, entacapone
MeSH Terms: conditions — Parkinson Disease | interventions — entacapone

INTERVENTIONS:
Drug: Entacapone

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the long-term treatment of entacapone in patients with Parkinson's disease with end-of-dose wearing-off.

This study is not recruiting patients in the United States.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of the long-term treatment of entacapone in patients with Parkinson's disease with end-of-dose wearing-off.

ELIGIBILITY:
Inclusion Criteria:

* Attended the Phase IIb study
* Able to fill out the patient diary

Exclusion Criteria:

* Serious heart, pulmonary, renal, hepatic or gastrointestinal disease
* Dementia symptoms
* Pregnant or nursing (lactating) women

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2003-02; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events during the long term treatment (maximum 3 years)
Blood pressure at every 12 weeks
Laboratory test at every 16 weeks
ECG at every 16 weeks

SECONDARY OUTCOMES:
On time based on patient diary (up to 104 weeks)
UPDRS score at every 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States